CLINICAL TRIAL: NCT06100640
Title: Paracervical Pouch Significance in Placenta Accreta Spectrum
Brief Title: Paracervical Pouch in Placenta Accreta Spectrum
Acronym: pouch
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Omar elshorbagy, lecturer in obstetrics and gynecology, faculty of medicine, Alexandria University
Other Study IDs: 26/564
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Placenta Accreta
Keywords: placenta adherence
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive paracervical pouch: The first group will include patients in whom a paracervical pouch is detected by transvaginal ultrasound.
- negative paracervical pouch: the second group will include patients in whom the pouch is not detected by transvaginal ultrasound

SUMMARY:
The study objective is the significance of the ultrasound detection of the paracervical pouch in placenta accreta spectrum. It aimed to evaluate its relation to the degree of placenta accreta spectrum, amount of the blood loss and the number of packed red blood cells transfused.

DETAILED DESCRIPTION:
The study will be carried on patients diagnosed with placenta previa or placenta accreta spectrum and had at least one caesarean section. The study will be divided into 2 groups of 70 patients at least per each. The first group will include patients in whom a paracervical pouch is detected, and the second group will include patients in whom the pouch is not detected by transvaginal ultrasound.

paracervical pouch is defined ultrasonographic as the downward displacement of the uterine serosa from the level of the cervical internal os

ELIGIBILITY:
Inclusion Criteria:

* • Patients between 19 to 40 years old

  * Patients had at least one cesarean section.

Exclusion Criteria:

* • Patients who request hysterectomy.

  * Patients diagnosed with hepatitis B, C, or HIV,
  * Those with bleeding diathesis.
  * Patients whose BMI is more than 40 kg/m2.
  * Patients who need an emergency cesarean section.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all patients who can be pregnant
Study Population: The study will be carried out on pregnant patients diagnosed with placenta previa or placenta accreta spectrum and who had at least one cesarean section. The study will be divided into 2 groups of 70 patients at least per each. The first group will include patients in whom a paracervical pouch is detected, and the second group will include patients in whom the pouch is not detected by transvaginal ultrasound.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
the rate of intraoperative diagnosis of placenta accreta spectrum | intraoperative
  the number of patients diagnosed intraoperatively with placenta accreta spectrum according to international federation of obstetrics and gynecology in both groups.
calculated amount of blood loss | intraoperative and 24 hours postoperative
  the total amount blood lost intraoperatively in millilitres.
blood transfusion | intraoperative and 24 hours postoperative
  the amount of packed red blood cell, fresh frozen plasma and platelets transfused in both groups.
rate of hysterectomy | intraoperative till 40 days postoperative
  the percentage of cases had hysterectomy in both groups.
internal iliac artery ligation | intraoperative
  the rate of internal iliac artery ligation in both groups.
Intensive care unit admission | postoperative for 5 days
  the number of patients admitted to the intensive care unit and the duration of their stay.
hospital stays | postoperative for 1 month
  the duration of hospital stays after the operation.
the presence of intraoperative pouch | intraoperative
  the detection of an intraoperative paracervical pouch grossly.

SECONDARY OUTCOMES:
total operation time | intraoperative
  the duration from the skin incision till skin closure.
repair time | intraoperative
  the duration from the placental separation till closure of the first layer.
preoperative hemoglobin levels in gm/dl | 24 hours before the operation
  the amount of the hemoglobin measured in gm/dl before the operation in both groups.
postoperative hemoglobin levels in gm/dl | 6 hours postoperative
  the amount of the hemoglobin measured in gm/dl after the operation in both groups.
rate of uterine wall disruption | intraoperative
  the number of patients who have a disruption of their anterior uterine wall during bladder dissection or placental separation in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
yes i would like to share the study protocol and the statistical analysis plan

REFERENCES:
- [Result] Shih JC, Kang J, Tsai SJ, Lee JK, Liu KL, Huang KY. The "rail sign": an ultrasound finding in placenta accreta spectrum indicating deep villous invasion and adverse outcomes. Am J Obstet Gynecol. 2021 Sep;225(3):292.e1-292.e17. doi: 10.1016/j.ajog.2021.03.018. Epub 2021 Mar 17. PMID 33744177